CLINICAL TRIAL: NCT04699331
Title: Individualized Brain Stimulation Using Transcranial Direct Current Stimulation Simulation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07-107
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized stimulation group (Experimental): Patients receive five sessions of individualized stimulation obtained from brain image-based transcranial direct stimulation simulation. The simulator generates the electrode's location on the scalp.
  Interventions: Device: Transcranial Direct Current Stimulation
- Conventional stimulation group (Active Comparator): Patients receive five sessions of conventional stimulation with electrodes over C3 and C4 based on the 10-20 system.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham stimulation group (Sham Comparator): Patients receive five sessions of sham stimulation with electrodes over C3 and C4 based on the 10-20 system.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation is a form of noninvasive neuromodulation that uses constant and low direct current delivered via electrodes on the scalp.

SUMMARY:
This study is to investigate the effect of transcranial direct current stimulation (tDCS) simulation-based individualized stimulation compared to conventional stimulation and sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke patients
* Chronic patients over 6 months after onset
* Patients with motor evoked potential of the first dorsal interosseous muscle
* Patients with the movement of fingers

Exclusion Criteria:

* History of psychiatric disease
* Significant other neurological diseases except for stroke
* Difficult to perform this experiment
* Patients who are deemed difficult to participate in this research by the investigator
* Patients with metal implants and medical devices
* History of epilepsy
* Pregnancy
* Skin defect at the site of electrode attachment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in motor evoked potential | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  Resting motor threshold (rMT), amplitude, and latency of motor evoked potential in the first dorsal interosseous muscle are measured. These outcomes are measured by transcranial magnetic stimulation over the motor hotspot. The rMT is defined as the minimum stimulus intensity that produced a minimal motor evoked response at rest. The amplitude means peak to peak of the muscle response. The latency is defined as the time point from the onset of the stimulus to the onset of MEP.

SECONDARY OUTCOMES:
Jebsen-Taylor hand function test | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  This test is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).
9-hole peg test | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Grip & Tip pinch strength test | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Box & Block test | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
Fugl-Meyer Assessment | Baseline, 1 day (immediately after one brain stimulation session) and about 14 days (immediately after five brain stimulation sessions)
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.
Sequential motor test | Baseline, 1 day (immediately after one brain stimulation session), 5 days (immediately before and after three brain stimulation sessions), and about 14 days (immediately before and after five brain stimulation sessions)
  Response time and accuracy are measured during finger tapping task.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea